CLINICAL TRIAL: NCT07027956
Title: A Comparison of Respiratory Function, Exercise Capacity and Oxygenation Between Smokers and Non-smokers
Brief Title: Respiratory Function and Oxygenation in Smokers and Non-smokers
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2025-08/88
Record Dates: First submitted 2025-05-28; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Smoking, Tobacco
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokers
- Non-smokers

SUMMARY:
This study aimed to compare respiratory function, exercise capacity, and intercostal muscle oxygenation in healthy smokers and non-smokers.

ELIGIBILITY:
Inclusion Criteria (Smokers):

* According to the World Health Organization and ICD smoking addiction criteria, consuming at least one cigarette every day for the last year
* Volunteering to participate in research
* Able to walk and cooperate

Exclusion Criteria (Smokers):

* Having any cardiopulmonary disease
* Having a musculoskeletal problem that could affect the tests
* Failure to comply with tests

Inclusion Criteria (Non-smokers):

* According to the World Health Organization and ICD smoking addiction criteria, having never smoked or not having smoked in the last year
* Volunteering to participate in research
* Able to walk and cooperate

Exclusion Criteria (Non-smokers):

* Having any cardiopulmonary disease
* Having a musculoskeletal problem that could affect the tests
* Failure to comply with tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with smokers and non-smokers will be included in the study.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity | 1st day
  Forced vital capacity (FVC) will be assessed using spirometry.
Forced expiratory volume in one second | 1st day
  Forced expiratory volume in one second (FEV1) will be assessed using spirometry
Forced expiratory volume in one second/forced vital capacity ratio | 1st day
  Forced expiratory volume in one second/forced vital capacity ratio will be assessed using spirometry.
Peak expiratory flow | 1st day
  Peak expiratory flow (PEF) will be assessed using spirometry.
Forced mid-expiratory flow | 1st day
  Forced mid-expiratory flow (FEF25-75) will be assessed using spirometry.
Inspiratory muscle strength | 1st day
  Strength index will be evaluated.
Exercise capacity | 2nd day
  will be evaluated with 6 minute walk test and total distance will be recorded.
Intercostal muscle oxygenation | 2nd day
  During the 6-minute walking test, oxygenation of the intercostal muscles will be evaluated with a monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)